CLINICAL TRIAL: NCT02012660
Title: Relationship Between Heat Wave and Moderate to Severe Hyponatremia in the Emergency Departement of Primary and Tertiary Care Teaching Hospital.
Brief Title: Relationship Between Heat Wave and Hyponatremia
Status: Completed | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Olivier T. Rutschmann, MD, University Hospital, Geneva
Other Study IDs: SU-051213
Record Dates: First submitted 2013-12-05; First posted 2013-12-16 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2015-04

CONDITIONS: Hyponatremia
MeSH Terms: conditions — Hyponatremia

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hyponatremia, seasonality: Summer months = June, July, August Winter months = December, January, February
  Interventions: Other: Seasonality

INTERVENTIONS:
Other: Seasonality — The impact of high temperature during summer months on the prevalence of hyponatremia will be explores.
  Other Names: Summer = June, July, August; Winter = December, January, February

SUMMARY:
The objective of this study is to explore the relationship between moderate to severe hyponatremia and heat.

DETAILED DESCRIPTION:
We will explore the relationship between heat wave and moderate and severe hyponatremia in a population of adult patients admitted in the emergency department of a primary and tertiary care teaching urban hospital. We will compare the prevalence of hyponatremia between summer and winter periods. We will describe the types of observed hyponatremia and describe the characteristics of the patients suffering of moderate to severe hyponatremia.

ELIGIBILITY:
Inclusion Criteria:

* all adults (> 16 y) with blood natremia measured

Exclusion Criteria:

* Patients without measure of natremia in the emergency department

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adults admitted to the emergency departement of a primary and tertiary care teaching hospital
Sampling Method: Non-Probability Sample
Enrollment: 28734 (Actual)
Dates: Start 2014-02; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Number of patients with moderate to severe hyponatremia | Natremia measured at admission in the ED
  Moderate to severe hyponatremia is defined as Sodium blood levels < 125 mmol/L

SECONDARY OUTCOMES:
Mortality | December 2011 to August 2013
Hospital length of stay | December 2011 to August 2013

CONTACTS AND LOCATIONS:
Overall Officials: Olivier T Rutschmann, MD, MPH, Principal Investigator — University Hospital, Geneva
Locations (1):
- Geneva University, Geneva, Canton of Geneva, Switzerland